CLINICAL TRIAL: NCT02228902
Title: Iron Absorption Trial
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rijnstate Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Ironabsorption
Record Dates: First submitted 2014-08-13; First posted 2014-08-29 (Estimated); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Iron Absorption; Bariatric Surgery; Roux- en -y Gastric Bypass
MeSH Terms: interventions — ferrous fumarate; ferrous gluconate

ARMS (2):
- ferrous fumarate (Active Comparator): 12 patients receive ferrous fumarate, 12 patients receive ferrous gluconate
  Interventions: Drug: Ferrous fumarate
- ferrous gluconate (Active Comparator): 12 patients receive ferrous fumarate and 12 patients receive ferrous gluconate
  Interventions: Drug: Ferrous gluconate

INTERVENTIONS:
Drug: Ferrous fumarate — one group receives ferrous fumarate (12 patients) and one group (12 patients) receives ferrous gluconate
  Arms: ferrous fumarate
Drug: Ferrous gluconate — One group receives ferrous fumarate and one group receives ferrous fumarate.
  Other Names: Losferron
  Arms: ferrous gluconate

SUMMARY:
Introduction: There are indications that the absorption of oral iron supplementation is reduced after a Roux- en -Y gastric bypass. Nevertheless, oral preparations are used as standard therapy for iron deficiency, even in patients who underwent a Roux- en -Y gastric bypass. Our goal is to evaluate if iron absorption is disturbed after a RYGB, which leads to a insufficient treatment of oral iron suppletion.

Methods: an iron absorption test will be performed pre- and postoperatively in 24 patients. Two groups will be created.

Preoperatively group 1 receives a daily dose of ferrous fumarate (600mg) and group 2 receives a daily dose Losferron (1390mg).

Before intake of the medicines, a fasting blood sample is taken (baseline), serum iron including ferritin, transferrin and transferrin saturation will be measured. After intake of losferron/ferrous fumarate blood samples will be taken 1, 2, 3, 4, 5 and 6 hours after intake, using a drip. An increase of 80 microgram/l is representative for a sufficient iron absorption. All patients undergo a Roux- en -Y gastric bypass.

Postoperatively; one month postoperatively the same absorption test will be repeated in the same patients.

ELIGIBILITY:
Inclusion Criteria:

* patients who are eligible for a primary Roux- en -Y gastric bypass and who have no pre-existing iron deficiency (serum ferritin between 20-200 micrograms/L)

Exclusion Criteria:

* blood transfusion one month before ans in the study period. The use of iron containing nutritional supplements, except our standardized multivitamin supplements. Decreased function of the kidney with a GFR of < 30ml/min and a serum creatinin below 50 micromol/L. Hb< 7.4 mmol/L in females en Hb< 8.4 mmol/L in males. Accumulation of iron. Hypersensitivity for ons of the medicinal products. Psychiatric illness. Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2015-05 (Actual); Study Completion 2015-05-04 (Actual)

PRIMARY OUTCOMES:
Iron values in the blood | 1 month after surgery
  Iron levels in teh blood will be measured before and 1,2,3,4,5 and 6 hours after the administration of oral iron replacement in micrograms / dl. This will take place before surgery and one month after surgery. The primary outcome is de difference between iron values pre- and postoperatively.

SECONDARY OUTCOMES:
difference in absorption between ferrous fumarate and ferrous gluconate | 1 month after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Rijnstate hospital, Arnhem, Netherlands

REFERENCES:
- [Derived] Schijns W, Ligthart MAP, Berends FJ, Janssen IMC, van Laarhoven CJHM, Aarts EO, de Boer H. Changes in Iron Absorption After Roux-en-Y Gastric Bypass. Obes Surg. 2018 Jun;28(6):1738-1744. doi: 10.1007/s11695-017-3088-5. PMID 29327182